CLINICAL TRIAL: NCT00100958
Title: Phase I Ascending Single Dose Pharmacokinetics (PK) and Safety Study of 3,3' Di-Indolymethane (DIM) Nutritional Product
Brief Title: Indole-3-Carbinol in Preventing Cancer in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000406002; KUMC-HSC-9139-2
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2006-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — indole-3-carbinol

INTERVENTIONS:
Drug: indole-3-carbinol

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of indole-3-carbinol may prevent cancer.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of indole-3-carbinol and to see how well it works compared to placebo in preventing cancer in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of indole-3-carbinol in healthy participants.
* Determine the safety and tolerability of this drug in these participants.
* Determine the pharmacokinetics of this drug in these participants.

Secondary

* Determine the effects of this drug on selected markers of sexual function in these participants.
* Determine the effects of this drug on markers of susceptibility to cancer in these participants.

OUTLINE: This is a randomized, double-blind, placebo-controlled, dose-escalation study. Participants at each dose level are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive a single dose of oral indole-3-carbinol on day 1.
* Arm II: Participants receive a single dose of oral placebo on day 1. Cohorts of 3 participants receive escalating doses of indole-3-carbinol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 participants experiences dose-limiting toxicity. An additional cohort of 3 participants is treated at the MTD.

Participants are followed on days 2, 3, and 6.

PROJECTED ACCRUAL: A total of 24 participants (18 in arm I and 6 in arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants

  * Non-smoker
  * No drug abuse, as determined by urine cotinine and baseline drug screen

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* Not specified

Life expectancy

* At least 12 months

Hematopoietic

* Absolute granulocyte count > 1,500/mm^3
* Hemoglobin > 10 g/dL

Hepatic

* Bilirubin < 1.8 mg/dL
* AST and ALT < 110 U/L
* Alkaline phosphatase < 300 U/L

Renal

* Creatinine < 2.0 mg/dL
* Albumin > 3.0 g/dL

Pulmonary

* No asthma

Other

* Not pregnant or nursing
* Negative pregnancy test
* Weight within 20% of ideal body weight by the Metropolitan Life table
* No serious drug allergies
* No arthritis
* No acute, unstable, chronic, or recurring medical condition
* No strict vegetarians
* No diabetes
* No evidence of an active malignancy
* No other serious intolerance or allergies

  * Mild seasonal allergies allowed
* No other serious acute or chronic illness
* None of the following chronic conditions:

  * Headaches
  * Dysphoria
  * Fatigue
  * Dizziness
  * Blurred vision
  * Insomnia
  * Rhinorrhea
  * Nausea
  * Vomiting
  * Abdominal pain
  * Diarrhea
  * Constipation
  * Premenstrual syndrome
* Cessation of menses within the past 10 days (menstruating women only)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Concurrent oral contraceptives allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 21 days since prior medications, herbal products, dietary supplements, or high-dose vitamins
* More than 3 months since prior investigational drugs
* At least 14 days since prior and no concurrent ingestion of cruciferous vegetables, including any of the following:

  * Broccoli
  * Cabbage, including coleslaw
  * Cauliflower
  * Bok-choy
  * Brussels sprouts
  * Collards
  * Kale
  * Kohlrabi
  * Mustard greens
  * Rutabaga
  * Turnip
  * Watercress
* At least 7 days since prior and no concurrent alcohol consumption
* At least 48 hours since prior ingestion of grapefruit-containing foods and beverages
* No concurrent chronic drug therapy
* No other concurrent supplements, including dietary supplements, vitamins, herbal products, or over-the-counter medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reed, PhD, Principal Investigator — University of Kansas
Locations (1):
- Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas, United States